CLINICAL TRIAL: NCT00368628
Title: Continuous Positive Airway Pressure for the Treatment of Acute Ischemic Stroke: A Feasibility Pilot Study
Brief Title: Continuous Positive Airway Pressure for the Treatment of Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Dawn M. Bravata, M.D., Roudebush VAMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0405026711
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-03

CONDITIONS: Acute Ischemic Stroke; Sleep Apnea
Keywords: acute ischemic stroke; sleep apnea; continuous positive airway pressure
MeSH Terms: conditions — Ischemic Stroke; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

INTERVENTIONS:
Procedure: continuous positive airway pressure — Continuous Positive Airway Pressure initiated within 48 hours of stroke onset and continued for 90 days.

SUMMARY:
New stroke therapies are needed. This study seeks to provide the preliminary data needed to plan a future study that will evaluate the efficacy of using continuous positive airway pressure (CPAP) to treat stroke patients who have sleep apnea. Our goal is to use this therapy to reduce stroke symptom severity.

DETAILED DESCRIPTION:
BACKGROUND Sleep apnea occurs in 60-96% of stroke survivors and is associated with poor functional recovery and higher post-stroke mortality. Among patients without stroke, continuous positive airway pressure (CPAP) is a safe and effective treatment for sleep apnea. This feasibility pilot study is a step in planning a future efficacy trial of CPAP for patients with acute ischemic stroke.

OBJECTIVES The primary objectives are, among acute ischemic stroke patients, to: (1) determine the feasibility of performing polysomnography; (2) refine the process for providing CPAP within 48-hours of stroke onset; and (3) determine the effect of CPAP on blood pressure.

METHODS This randomized controlled feasibility study will enroll 100 acute ischemic stroke patients. Intervention patients (N=60) receive CPAP within 48 hours of stroke onset and continuing for up to 30 days. At 30 days post-enrollment, the intervention patients undergo unattended polysomnography. Control (N=40) patients receive unattended polysomnography at baseline and after 30 days.

SIGNIFICANCE CPAP represents an important new potential therapy for acute stroke. CPAP may reduce both the neurological symptom severity of the acute stroke and prevent stroke recurrence.

ELIGIBILITY:
Inclusion Criteria: acute ischemic stroke with NIH Stroke Scale >=2 -

Exclusion Criteria: respiratory distress; COPD requiring oxygen; primary intracranial hemorrhage on admission brain imaging; time from symptom onset to sleep study or CPAP treatment >72 hours or time from hospital admission to sleep study or CPAP treatment >48 hours; life expectancy less than 6 months; inability to provide informed consent; inability to communicate in English; residence outside the greater New Haven area; or any condition where the monitoring required by the study would constitute a risk to the patient or impair his or her care.

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
proportion using CPAP within 48-hours of stroke onset | 72 hours

SECONDARY OUTCOMES:
prevalence of sleep apnea | 30 days post stroke

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M Bravata, MD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Bravata DM, Concato J, Fried T, Ranjbar N, Sadarangani T, McClain V, Struve F, Zygmunt L, Knight HJ, Lo A, Richerson GB, Gorman M, Williams LS, Brass LM, Agostini J, Mohsenin V, Roux F, Yaggi HK. Continuous positive airway pressure: evaluation of a novel therapy for patients with acute ischemic stroke. Sleep. 2011 Sep 1;34(9):1271-7. doi: 10.5665/SLEEP.1254. PMID 21886365